CLINICAL TRIAL: NCT03271216
Title: Surveillance Monitoring on General Wards
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00066847
Record Dates: First submitted 2015-04-08; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: No intervention — no intervention

SUMMARY:
This is a study to determine if surveillance monitoring of general ward patients can reduce cardio-pulmonary arrest while maintaining an acceptable false alarms rate for nursing workload.

DETAILED DESCRIPTION:
The investigators placed a wired monitoring system (pulse oximetry, heart rate and respiratory rate) on every patient who arrived on a subject general post surgical ward who assented to wear the system. this was the Masimo PSNET system using the Radical 87 monitor and an acoustic respiratory sensor along with a Masimo pulse oximetry probe. Patients were monitored for a minimum of 48 hrs. Heart Rate (HR) parameters were set between 45-130, Respiratory rate was set between 6-20 and pulse oximetrry was 85-100%. Nurses documented in the Electronic Medical Record (EMR) any alarms they responded to as to whether they were false (vital sign not out of range when rechecked) or true and what the response was. Responses ranged from nurse managed to notification of primary service to Rapid Response Activation to Code team activation as well as transfer to a higher level of care (operating room or Intensive Care Unit (ICU)/IMC. Patient and Nursing satisfaction surveys were collected.

ELIGIBILITY:
Inclusion Criteria:

* all post-surgical patients admitted to a post-operative general hospital ward

Exclusion Criteria:

* inability to understand English or provide verbal consent for data analysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-surgical patients on a general hospital ward
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
positive predictive value (PPV) | 6 months
  The PPV of the wired monitoring system (pulse oximetry, heart rate and respiratory rate) will be determined based on change in vital signs (HR<45 or >130, RR<6 or >20 and pulse oximetry <85) indicating clinical deterioration